CLINICAL TRIAL: NCT04016519
Title: Evaluation of the Quality of Life of the Caregivers Following the Installation of a Gastrostomy in the Child
Brief Title: The Quality of Life of Children With Gastrostomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-66; RC18_0352 (Registry Identifier: APHM)
Record Dates: First submitted 2019-06-18; First posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Gastrostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastrostomie: Gastrostomy involves creating an opening between the skin and the stomach. It allows the administration of nutrition solutes or food directly into the stomach without passing through the mouth and esophagus. It is a method widely used since the 1980s for enteral nutrition.
  In the field of pediatrics, gastrostomy is considered in chronic diseases when enteral nutrition is necessary in the long term.
  Interventions: Other: Gastrostomie

INTERVENTIONS:
Other: Gastrostomie — Gastrostomy involves creating an opening between the skin and the stomach. It allows the administration of nutrition solutes or food directly into the stomach without passing through the mouth and esophagus. It is a method widely used since the 1980s for enteral nutrition.
  In the field of pediatrics, gastrostomy is considered in chronic diseases when enteral nutrition is necessary in the long term.

SUMMARY:
Study the quality of life with generic questionnaires (17-20), validated and used in other pathologies and chronic diseases of the child. This will allow reproducibility and comparisons to other populations, general or other chronic diseases (acute leukemias ...). This is to conduct a pilot study, preliminary to the construction of a larger study, longitudinal with several evaluation times.

DETAILED DESCRIPTION:
Gastrostomy involves creating an opening between the skin and the stomach. It allows the administration of nutrition solutes or food directly into the stomach without passing through the mouth and esophagus. It is a method widely used since the 1980s for enteral nutrition.

In the field of pediatrics, gastrostomy is considered in chronic diseases when enteral nutrition is necessary in the long term. The percutaneous endoscopic method is nowadays one of the most widespread methods that has proven effective on growth and nutrition, with few side effects. Few studies have analyzed children's quality of life after gastrostomy. On the one hand, it increases the perceived health after the pose. It allows a reduction of the stress of the parents, at a distance from the pose, and its insertion would be chosen again by the parents if it were to do again. Meals and medication administration would be easier for parents with a decrease in frequency and time for meals. But on the other hand, its insertion is often difficult for families to experience by changing the diet. The family dynamics is modified and it would lead to logistical constraints for meals or outings . The vision of the corporal schema would also be altered. Following a systematic review of the literature conducted in early 2018, there are currently only 12 cross-sectional studies assessing the quality of life of caregivers after gastrostomy . The numbers vary from 24 to 100 with an average of 65. The results of these studies are generally positive with an improvement in the quality of life and a high degree of satisfaction of carers.

These studies reveal logistical difficulties for social contacts and meals as well as for the re-education of their child. They also raise a lack of information on the part of health professionals. These studies were conducted with different, non-standardized self-questionnaires. None of these studies conducted a direct assessment of the child using a questionnaire designed for them. This assessment of children can be performed in children of understanding age and having a pathology that allows them to communicate. It allows an approach and a direct vision of the quality of life. The investigator's goal is to study the quality of life with generic questionnaires, validated and used in other pathologies and chronic diseases of the child. This will allow reproducibility and comparisons to other populations, general or other chronic diseases (acute leukemias ...). This is to conduct a pilot study, preliminary to the construction of a larger study, longitudinal with several evaluation times.

ELIGIBILITY:
Inclusion Criteria:

Child:

* 1 month to 17 years old;
* Not opposed to participating in the study;
* Whose parent or legal representative did not object to participating in the study;
* Having a pathology requiring enteral nutrition in the long term exclusive or mixed;
* Having had a gastrostomy between January 2014 and 2019.

Helping :

* Be the parent or legal representative of the child who meets the criteria for inclusion and non inclusion;
* Not opposed to participating in the study;
* Having the ability to comply with the protocol requirements (in particular: understanding and speaking French).

Exclusion Criteria:

Child:

* Refusing to participate in the study;
* Child who has died or no longer has gastrostomy.

Helping :

* Inability to comply with study protocol, or investigator uncertainty about willingness or ability to comply with protocol requirements;
* Refusing to participate in the study

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and caregivers with gastronomy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the body mass index | 10 Months
  Observation of a decrease in body mass index for patient with gastrostomy

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France